CLINICAL TRIAL: NCT00001390
Title: Salivary Evaluation in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940018; 94-D-0018
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09-20

CONDITIONS: Healthy; Salivary Gland Disease
Keywords: Saliva; Parotid; Lip Biopsy; Health; Exocrine; Normal Volunteer
MeSH Terms: conditions — Salivary Gland Diseases

SUMMARY:
Saliva is critical in maintaining oral health and comfort. Our laboratory has investigated several disorders of salivary glands. The purpose of this protocol is to obtain data from healthy volunteers for comparison with data from patients with salivary dysfunction. We plan to utilize the NIH Clinical Center Clinical Research Volunteer Program to solicit paid participation from healthy adults. Study procedures are accomplished in 2-3 outpatient visits that include an interview, saliva collection, lip biopsy, clinical laboratory studies, dry eye examination, and lip biopsy follow up, as needed. These are routine diagnostic procedures. Biopsy specimens may be used in clinical and laboratory studies, such as in vitro biochemical analysis or in vivo transplantation.

Some of the Healthy Volunteers may be asked to participate in an MRI study of the salivary glands.

DETAILED DESCRIPTION:
* Objective: To obtain data from healthy volunteers for comparison with data from patients with salivary dysfunction.
* Study population: Healthy volunteers aged 18-70 years old
* Design: Observational
* Outcome measures: Clinical and basic science data to serve as controls for comparisons with subjects presenting with salivary gland dysfunction

Saliva is critical in maintaining oral health and comfort. Our laboratory has investigated several disorders of salivary glands. The purpose of this protocol is to obtain data from healthy volunteers for comparison with data from patients with salivary dysfunction. We plan to utilize the NIH Clinical Center Clinical Research Volunteer Program to solicit paid participation from healthy adults. Study procedures are accomplished in 2-3 outpatient visits that include an interview, saliva collection, lip biopsy, clinical laboratory studies, dry eye examination, and lip biopsy follow up, as needed. These are routine diagnostic procedures. Biopsy specimens may be used in clinical and laboratory studies, such as in vitro biochemical analysis or in vivo transplantation.

Some of the Healthy Volunteers may be asked to participate in an MRI study of the salivary glands.

The outcome measurement for this study is to determine those healthy subjects whose data and specimens can be used as control comparison for our patient subjects in our Sj(SqrRoot)(Delta)gren s syndrome studies (15-D-0051, 99-D-0070, 11-D-0094 and/or 11-D-0172).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Healthy male or female volunteers from 18 to 70 years old.
* Ability to understand and sign an informed consent document.

EXCLUSION CRITERIA:

* Known pregnancy.
* Chronic medical illness, other than well-controlled hypertension or hyperlipidemia.
* Chronic use of medications, with the exception of oral contraceptives, hormone replacement therapy, antihypertensives and antilipemics.
* Have problems with dry mouth and/or dry eyes.
* NIH employees who are subordinates/relatives/co-workers of investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 1993-10-26; Study Completion 2018-09-20

CONTACTS AND LOCATIONS:
Overall Officials: Blake M Warner, D.D.S., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Tanaka T, Warner BM, Odani T, Ji Y, Mo YQ, Nakamura H, Jang SI, Yin H, Michael DG, Hirata N, Suizu F, Ishigaki S, Oliveira FR, Motta ACF, Ribeiro-Silva A, Rocha EM, Atsumi T, Noguchi M, Chiorini JA. LAMP3 induces apoptosis and autoantigen release in Sjogren's syndrome patients. Sci Rep. 2020 Sep 16;10(1):15169. doi: 10.1038/s41598-020-71669-5. PMID 32939030
- [Derived] Burbelo PD, Ferre EMN, Chaturvedi A, Chiorini JA, Alevizos I, Lionakis MS, Warner BM. Profiling Autoantibodies against Salivary Proteins in Sicca Conditions. J Dent Res. 2019 Jul;98(7):772-778. doi: 10.1177/0022034519850564. Epub 2019 May 16. PMID 31095438
- [Derived] Yin H, Cabrera-Perez J, Lai Z, Michael D, Weller M, Swaim WD, Liu X, Catalan MA, Rocha EM, Ismail N, Afione S, Rana NA, Di Pasquale G, Alevizos I, Ambudkar I, Illei GG, Chiorini JA. Association of bone morphogenetic protein 6 with exocrine gland dysfunction in patients with Sjogren's syndrome and in mice. Arthritis Rheum. 2013 Dec;65(12):3228-38. doi: 10.1002/art.38123. PMID 23982860